CLINICAL TRIAL: NCT01275274
Title: Retinoids in ANCA Small Vessel Vasculitis: Silencing Autoantigens
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no subject enrolled in nearly 2 years
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-2007; P01DK058335 (NIH)
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-09

CONDITIONS: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis
Keywords: ANCA; Vasculitis; Pauci-immune vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis | interventions — Tretinoin; Standard of Care; Azathioprine; Adenosine Triphosphate; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (Active Comparator): maintenance therapy with azathioprine or mycophenolate mofetil with or without small dose prednisone.
  Interventions: Drug: Standard of care
- Retinoic acid (Experimental): Tretinoin in addition to standard of care
  Interventions: Drug: Retinoic acid

INTERVENTIONS:
Drug: Retinoic acid — Patients will be started at half the recommended dose of retinoic acid for the treatment of acute promyelocytic leukemia (APL), i.e. 22.5mg/m2/day orally in two divided doses, to minimize the risk of adverse events. If there is no decrease in PR3/MPO gene expression to a fold change of < 2 by quantitative polymerase chain reaction(QT-PCR) technique for PR3 at the end of 4 weeks, the dose will be increased to 45 mg/m2/day in two divided doses for an additional 8 weeks. If the patient shows a decrease in PR3/MPO gene expression to < 2 at 4 weeks, the patient will remain on the same dose for the remainder of 12 weeks. All patients will be followed for a total of 12 months for safety evaluations and to assess changes in disease activity and the incidence of disease relapse.
  Other Names: Tretinoin
  Arms: Retinoic acid
Drug: Standard of care — maintenance therapy with azathioprine or mycophenolate mofetil with or without small dose prednisone. Dose, frequency and duration depend on disease activity (partial or complete remission).
  Other Names: Imuran, Azasan; Cellcept
  Arms: Standard of care

SUMMARY:
The purpose of this research study is to learn if adding all-trans retinoic acid (tretinoin) to conventional treatment of Anti- Neutrophil Cytoplasmic Autoantibodies (ANCA) vasculitis can decrease the level of disease activity.

DETAILED DESCRIPTION:
Neutrophils are white blood cells that are the target of the ANCA antibodies. T cells are white blood cells that are involved in regulating the immune system. Laboratory research studies suggest that all-trans retinoic acid (tretinoin) can affect the neutrophils and the T lymphocytes in such a way that could decrease the abnormal immune response directed against the body own neutrophils.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ANCA disease and no more than mild activity as determined by a BVAS score of 1 to 4. These are patients who will have undergone induction with cyclophosphamide and corticosteroids in the past, and will be in partial remission on maintenance therapy with azathioprine or mycophenolate mofetil with or without small dose prednisone. We anticipated that most patients enrolled in the study will have low grade persistent ("grumbling") disease on stable immunosuppressants.
* Documented 6-fold or greater elevation in PR3 and/or MPO gene expression by the RT-PCR technique. We estimate that approximately 25% of patients with a BVAS <5 will have an elevation in PR3 and/or MPO gene expression based on our previous studies. 2 Patients must be on stable maintenance therapy with prednisone (<10 mg/day or equivalent), cyclosporine A, mycophenolate mofetil or azathioprine for at least 8 weeks.

Exclusion Criteria:

* Patients with severe, active vasculitis requiring institution or an increase in dose of corticosteroids, cyclophosphamide, azathioprine, mycophenolate mofetil or any new immunosuppressive medication within the previous 8 weeks or at the time of enrollment.
* Pregnancy, breastfeeding, or unwillingness to use at least two contraceptive methods (at least one of which must be primary, including tubal ligation, partner vasectomy, oral contraceptives, implanted contraceptives, and intrauterine device). The rationale is that retinoids are teratogenic and are excreted in breast milk. Contraceptive methods must be instituted at least 1 month before starting tretinoin and continued at least 1 month after stopping the medication.
* History of hepatitis, cirrhosis or abnormal liver tests, including aspartate aminotransferase (AST), alanine aminotransferase (ALT), Alkaline phosphatase, Gamma-glutamyl transpeptidase (GGT), total bilirubin, or prothrombin time; unless the abnormality is due to a specific hepatotoxic medication, AND the liver test levels are l< 2 times the upper limit of the normal AND normalize upon holding the offending drug.
* Hypertriglyceridemia (>500 mg/dL) despite statin/fibrate therapy.
* Any medical conditions requiring concurrent use of tetracycline, minocycline, or doxycycline, due to enhanced risk of increased intracranial pressure.
* Any medical conditions requiring concurrent use of rifampin, phenobarbital, pentobarbital, ketoconazole, cimetidine, erythromycin, verapamil, diltiazem, vitamin A and antithrombotic agents (Tranexamic Acid, Aminocaproic Acid or Aprotinin)due to the potential for interactions with tretinoin therapy.
* Presence of unstable cardiovascular disease, uncontrolled diabetes with hemoglobin A1c > 8% g/dL, or chronic inflammatory or infectious conditions.
* Glomerular Filtration Rate (GFR) <25 ml/min/1.73m^2 as estimated by the MDRD equation, as the metabolites of retinoids are excreted in part in urine, and there is a concern for increased toxicity.
* Untreated depression, as retinoids have been associated with depression, suicidal ideation, and aggressive behavior.
* Neutropenia (neutrophil count < 1000 cell/mm^3).
* Known osteoporosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
change in leukocyte Myeloperoxidase (MPO) and Proteinase 3 (PR3) message | week 12
  normalization of PR3 and MPO message at the end of treatment.

SECONDARY OUTCOMES:
Birmingham Vasculitis Activity Score (BVAS) | 52 weeks
  (1) Change in BVAS at the end of treatment (week 12) and at week 52, compared to baseline (day 1); (2) Change in Treg and Th17 cells at weeks 12 and 52, compared to baseline (day 1); and (3) the frequency of relapse during the follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick H Nachman, MD, Principal Investigator — UNC Kidney Center
Locations (1):
- UNC Kidney Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
no data obtained.